CLINICAL TRIAL: NCT03900429
Title: A Phase 3, Multinational, Double-Blind, Randomized, Placebo-Controlled Study of MGL-3196 (Resmetirom) in Patients With Non-Alcoholic Steatohepatitis (NASH) and Fibrosis to Resolve NASH and Reduce Progression to Cirrhosis and/or Hepatic Decompensation
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of MGL-3196 (Resmetirom) in Patients With NASH and Fibrosis
Acronym: MAESTRO-NASH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGL-3196-11
Record Dates: First submitted 2019-03-26; First posted 2019-04-03 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — resmetirom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Matching Placebo (Placebo Comparator): Placebo Daily
  Interventions: Drug: Placebo; Procedure: Liver Biopsy
- 80 mg MGL-3196 (Active Comparator): 80 mg daily
  Interventions: Drug: MGL-3196; Procedure: Liver Biopsy
- 100 mg MGL-3196 (Active Comparator): 100 mg daily
  Interventions: Drug: MGL-3196; Procedure: Liver Biopsy

INTERVENTIONS:
Drug: MGL-3196 — Tablet
  Other Names: Resmetirom
  Arms: 100 mg MGL-3196; 80 mg MGL-3196
Drug: Placebo — Matching Tablets
  Arms: Matching Placebo
Procedure: Liver Biopsy — A procedure in which a needle is inserted into the liver to collect a tissue sample

SUMMARY:
A double-blind placebo controlled randomized Phase 3 study to determine if 80 or 100 mg of MGL-3196 as compared with placebo resolves NASH and/or reduces fibrosis on liver biopsy and prevents progression to cirrhosis and/or advanced liver disease

DETAILED DESCRIPTION:
Primary and secondary endpoint population at Week 52 will be at least 900 patients, more than half fibrosis score 3 (F3), the remainder fibrosis score 2 (F2) and <10% fibrosis score F1B (F1B) based on final liver biopsy baseline fibrosis score.

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing to participate in the study and provide written informed consent.
2. Male and female adults ≥ 18 years of age.
3. Suspected or confirmed diagnosis of NASH fibrosis suggested by the historical data. Meet one of the following criteria that is consistent with NASH liver fibrosis:

   1. Historical biochemical test for fibrosis: PRO-C3 >14 ng/mL or ELF ≥9
   2. FibroScan with transient elastography ≥8.5 kPa and controlled attenuation parameter ≥280 dB.m-1
   3. Historical liver biopsy obtained <2 years before expected randomization showing Stage 1B, 2 or 3 fibrosis with NASH based on existing pathology review, with no significant change in body weight >5% or medication that might affect NAS or fibrosis stage.
4. MRI-PDFF fat fraction ≥8% obtained during the screening period
5. Biopsy-proven NASH (baseline liver biopsy) based on a liver biopsy obtained ≤6 months before anticipated date of randomization (if the biopsy is deemed acceptable for interpretation by the central reader) with fibrosis stage 1A/1C, 1B, 2, or 3 on liver biopsy and NAS of ≥4 with a score of at least 1 in each of the following NAS components:

   1. Steatosis (scored 0 to 3)
   2. Ballooning degeneration (scored 0 to 2)
   3. Lobular inflammation (scored 0 to 3)

Exclusion Criteria:

1. History of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to Screening.
2. Regular use of drugs historically associated with NAFLD
3. Thyroid diseases:

   1. Active hyperthyroidism.
   2. Untreated clinical hypothyroidism defined by thyroid stimulating hormone (TSH) >7 IU/L with symptoms of hypothyroidism or >10 IU/L without symptoms.
   3. Patients who have had a thyroidectomy and are on replacement thyroxine doses >75 µg per day are allowed.
4. History of bariatric surgery or intestinal bypass surgery within the 5 years prior to randomization or planned during the conduct of the study.
5. Recent significant weight gain or loss
6. HbA1c ≥ 9.0%.
7. Glucagon-like peptide 1 [GLP-1] agonist, high dose Vitamin E (> 400 IU/day), or pioglitazone therapy unless stable dose for 24 weeks prior to biopsy.
8. Presence of cirrhosis on liver biopsy defined as stage 4 fibrosis.
9. Diagnosis of hepatocellular carcinoma (HCC).
10. MELD score ≥12, as determined at Screening, unless due to therapeutic anti coagulation.
11. Hepatic decompensation
12. Chronic liver diseases other than NASH
13. Active autoimmune disease
14. Serum ALT > 250 U/L.
15. Active, serious medical disease with a likely life expectancy < 2 years.
16. Participation in an investigational new drug trial in the 60 days or 5 half-lives, whichever is longer.
17. Any other condition which, in the opinion of the Investigator, would impede compliance, hinder completion of the study, compromise the well-being of the patient, or interfere with the study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1759 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Week 52 Dual Primary Objectives: To determine the effect of 80 or 100 mg MGL-3196 vs matching placebo on liver biopsy (NASH CRN score) at Week 52 compared with Baseline | 52 weeks
  1. Proportion with resolution of NASH (ballooning 0, inflammation 0,1) associated with at least 2-point reduction in NAFLD Activity Score (NAS) without worsening of fibrosis stage OR
  2. Proportion with at least a 1-point improvement in fibrosis stage with no worsening of NAS
Month 54 Primary Objective: Time to experiencing an adjudicated Composite Clinical Outcome event (Final Primary Endpoint, at 54 months) | up to 54 months
  The Composite Clinical Outcome is composed of all-cause mortality, liver transplant, and significant hepatic events (including hepatic decompensation events [ascites, encephalopathy, or gastroesophageal variceal hemorrhage], histological progression to cirrhosis, and a confirmed increase of MELD score from <12 to ≥15).

SECONDARY OUTCOMES:
Week 52 Key Secondary Objective: To determine the effect of once-daily, oral administration of MGL-3196 80 or 100 mg versus matching placebo on the percent change from Baseline at 24 weeks in directly measured low-density lipoprotein cholesterol (LDL-C) | 24 weeks
  Assess the effect of MGL-3196 80 mg or 100 mg compared to placebo on LDL-C measured by percent change from Baseline at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Taub, MD, Study Director — Madrigal Pharmaceuticals, Inc.
Locations (246):
- United States (89):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - East Valley Family Physicians, Chandler, Arizona
  - The Institute for Liver Health - Chandler, Chandler, Arizona
  - The Institute for Liver Health - Glendale, Glendale, Arizona
  - Desert Clinical Research, Mesa, Arizona
  - Adobe Gastroenterology, Tucson, Arizona
  - The Institute for Liver Health - Tucson, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Fresno Clinical Research Center, Fresno, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - University of California San Diego, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - National Research Institute - Los Angeles, Los Angeles, California
  - Ruane Clinical Research, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - National Research Institute - Panorama City, Panorama City, California
  - Alliance Clinical Research, Poway, California
  - San Fernando Valley Health Institute, Van Nuys, California
  - Colorado Springs Family Practice, Colorado Springs, Colorado
  - South Denver Gastroenterology - Swedish Medical Center Office, Englewood, Colorado
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Covenant Metabolic Specialists - Fort Myers, Fort Myers, Florida
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami, Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Bioclinica Research - Orlando, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Research, Sarasota, Florida
  - Bioclinica Research - The Villages, The Villages, Florida
  - GI Specialists of Georgia, Marietta, Georgia
  - Clinical Research - Chicago, Chicago, Illinois
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Fairway, Kansas
  - Kansas Medical Clinic - Gastroenterology, Topeka, Kansas
  - Texas Digestive Disease Consultants - Gastroenterology Associates - Baton Rouge, Baton Rouge, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Clinical Trials of America, West Monroe, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Gastrointestinal Associates and Endoscopy Center - Madison, Flowood, Mississippi
  - Southern Therapy and Advanced Research, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Clinical Research US - Henderson, Henderson, Nevada
  - Mt. Sinai Medical Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - University of North Carolina Medical Center - Chapel Hill, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Lucas Research, Morehead City, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Aventiv Research - Columbus, Columbus, Ohio
  - Awasty Research Network, Marion, Ohio
  - Premier Medical Group - Clarksville, Clarksville, Tennessee
  - Gastro One - Germantown - Centre Oak Way, Germantown, Tennessee
  - Associates in Gastroenterology, Hermitage, Tennessee
  - Gastrointestinal Associates - Knoxville, Knoxville, Tennessee
  - South Texas Research Institute - Brownsville, Brownsville, Texas
  - Dallas Research Center, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Digestive Disease Consultants - Fort Worth, Fort Worth, Texas
  - Liver Associates of Texas, Houston, Texas
  - Doctor's Hospital at Renaissance, McAllen, Texas
  - Plano Research Center, Plano, Texas
  - Pinnacle Clinical Research - Austin, Rollingwood, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - San Antonio Research Center, San Antonio, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - Impact Research Institute, Waco, Texas
  - Texas Digestive Disease Consultants - Bay Area Gastroenterology, Webster, Texas
  - Wasatch Peak Family Practice, Layton, Utah
  - Salt Lake City Research Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Richmond, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Australia (14):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Saint Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Misericordiae, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (7):
  - Klinikum Klagenfurt Am Wörthersee, Klagenfurt, Carinthia
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz, Upper Austria
  - Krankenanstalt Rudolfstiftung, Vienna, Vienna
  - Landesklinik St. Veit, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (11):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - Hôpital Erasme, Brussels, Brussels Capital
  - Universitair Ziekenhuis Leuven, Leuven, Flemish Brabant
  - Ziekenhuis Oost-Limburg', Genk, Limburg
  - Algemeen Ziekenhuis Maria Middelares, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - AZ Delta Campus Wilgenstraat, Roeselare, West-Vlaanderen
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Universitaire Brugmann, Laken
  - Universitair Ziekenhuis Leuven, Leuven
- Canada (10):
  - University of Calgary Liver Unit, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - South Shore Medical Arts, Bridgewater, Nova Scotia
  - LMC/ Manna Research - Brampton, Brampton, Ontario
  - William Osler Health System, Brampton, Ontario
  - McMaster University, Hamilton, Ontario
  - Toronto General Hospital - Clinical Trials Pharmacy, Toronto, Ontario
  - Toronto Liver Center, Toronto, Ontario
  - Lair Centre, Vancouver
  - GI Research Institute, Vancouver
- France (19):
  - Les Hôpitaux Universitaires de Strasbourg - Hôpital Hautepierre, Strasbourg, Alsace
  - Nouvel Hôpital Civil, Strasbourg, Alsace
  - Hôpital de la Croix Rousse, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand, Auvergne
  - Centre Hospitalier Universitaire de Rennes, Rennes, Brittany Region
  - Hôpital Jean-Minjoz, Besançon, Franche-Comte
  - Centre Hospitalier Régional Universitaire de Lille, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Montpellier, Montpellier, Languedoc-Roussillon
  - Hôpital Dupuytren, Limoges, Limousin
  - Centre Hospitalier Universitaire de Toulouse - Hôpital Rangueil, Toulouse, Midi-Pyrenees
  - Center Hospitalier Universitaire d'Angers, Angers, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Nice Hôpital l'Archet, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Universitaire Amiens-Picardie, Amiens
  - Hôpital Beaujon, Clichy
  - Hôpital Universitaire Pitié Salpêtrière, Paris
  - Centre Hospitalier Universitaire de Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
  - Hôpital Avicenne, Bobigny, Île-de-France Region
  - Centre Hospitalier Universitaire Henri Mondor, Créteil, Île-de-France Region
  - Assistance Publique-Hôpitaux de Paris Hôpital Cochin, Paris, Île-de-France Region
- Germany (13):
  - Berlin Clinical Research Center, Berlin
  - Charité Universitätsmedizin Berlin - Campus Mitte, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - EPIMED, Berlin
  - Zentrum für Infektiologie Berlin Prenzlauer Berg, Berlin
  - Frankfurt Clinical Research Center, Frankfurt am Main
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum des Saarlandes, Homburg
  - EUGASTRO, Leipzig
  - Leipzig Research Center, Leipzig
  - SIBAmed Studienzentrum, Leipzig
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (7):
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház, Békéscsaba, Bekes County
  - Magyarország Egészségügyi Szolgáltató - Gyula, Gyula, Bekes County
  - Debreceni Egyetem Kenézy Gyula Egyetemi Kórház, Debrecen, Hajdú-Bihar
  - Magyarország Research Center, Debrecen, Hajdú-Bihar
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet, Budapest
  - Magyarország Research Center, Budapest
- Israel (11):
  - The Chaim Sheba Medical Center, Ramat Gan, Tel Aviv
  - Emek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus - Rambam Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Western Galilee Hospital-Nahariya, Nahariya
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (12):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria Policlinico Gaetano Martino, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Polo Universitario - L'Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliera Universitaria-Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione (ISMETT), Palermo
  - Azienda Ospedaliero-Universitaria Pisana Ospedale Cisanello, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Universita degli Studi di Roma La Sapienza - Umberto I Policlinico di Roma, Roma
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Mexico (5):
  - Centro Integral en Reumatología, Guadalajara, Jalisco
  - Centro Mexicano de Desarrollo de Estudios Clínicos, Mexico City, Mexico City
  - Centro de Investigacion y Gastroenterologia, Mexico City, Mexico City
  - JM Research, Cuernavaca, Morelos
  - Investigaciones Médicas Cisneros, Monterrey, Nuevo León
- Poland (9):
  - Polska Oddział w Częstochowie, Częstochowa
  - Polska Oddział w Gdansk, Gdansk
  - Polska Oddział w Gdyni, Gdynia
  - Polska Oddział w Katowicach, Katowice
  - Polska Oddział w Łodz, Lodz
  - Polska Oddział w Poznaniu, Poznan
  - Centrum Medyczne Pratia Poznan, Skórzewo
  - Polska Oddział w Warszawie, Warsaw
  - Polska Oddział w Wrocław, Wroclaw
- Fundación De Investigación De Diego, San Juan, Puerto Rico
- Spain (12):
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Consorci Hospital General Universitari de València, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Switzerland (3):
  - Universitatsspital Bern, Bern
  - Fondazione Epatocentro Ticino, Lugano
  - Universitatsspital Zurich, Zurich
- United Kingdom (23):
  - Midlands Clinical Research Centre, Birmingham, England
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Lancashire Clinical Research Centre, Chorley, England
  - North Teesside Clinical Research Centre, Hardwick, England
  - Merseyside Clinical Research Centre, Liverpool, England
  - Barts Health NHS Trust, London, England
  - Chelsea and Westminster Hospital NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust, London, England
  - Royal Free London NHS Foundation Trust, London, England
  - Manchester Clinical Research Centre, Manchester, England
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - Thames Valley Dedicated Research Centre, Reading, England
  - Belfast Health and Social Care Trust, Belfast, Northern Ireland
  - The Hexham Clinic, Hexham, Northumberland, England
  - The Wales Clinic, Cardiff, Wales
  - Abertawe Bro Morgannwg University Health Board, Swansea, Wales
  - Aintree University Hospitals NHS Foundation Trust, Liverpool
  - Saint George's University Hospitals NHS Foundation Trust, London
  - Plymouth Hospitals NHS Trust, Plymouth
  - Portsmouth Hospitals NHS Trust, Portsmouth

REFERENCES:
- [Derived] Noureddin M, Rinella M, Taub R, Labriola D, Camacho RC, Alkhouri N, Loomba R, Bansal MB. Effects of Resmetirom on Metabolic-Dysfunction Associated Steatohepatitis in Patients With Weight Loss and/or Diabetes Taking Glucagon-Like Peptide-1 Receptor Agonists and Other Diabetes Therapies: A Secondary Analysis of the MAESTRO-NASH Trial. Aliment Pharmacol Ther. 2025 Dec;62(11-12):1089-1099. doi: 10.1111/apt.70382. Epub 2025 Oct 23. PMID 41127972
- [Derived] Harrison SA, Bedossa P, Guy CD, Schattenberg JM, Loomba R, Taub R, Labriola D, Moussa SE, Neff GW, Rinella ME, Anstee QM, Abdelmalek MF, Younossi Z, Baum SJ, Francque S, Charlton MR, Newsome PN, Lanthier N, Schiefke I, Mangia A, Pericas JM, Patil R, Sanyal AJ, Noureddin M, Bansal MB, Alkhouri N, Castera L, Rudraraju M, Ratziu V; MAESTRO-NASH Investigators. A Phase 3, Randomized, Controlled Trial of Resmetirom in NASH with Liver Fibrosis. N Engl J Med. 2024 Feb 8;390(6):497-509. doi: 10.1056/NEJMoa2309000. PMID 38324483
- [Derived] Harrison SA, Ratziu V, Anstee QM, Noureddin M, Sanyal AJ, Schattenberg JM, Bedossa P, Bashir MR, Schneider D, Taub R, Bansal M, Kowdley KV, Younossi ZM, Loomba R. Design of the phase 3 MAESTRO clinical program to evaluate resmetirom for the treatment of nonalcoholic steatohepatitis. Aliment Pharmacol Ther. 2024 Jan;59(1):51-63. doi: 10.1111/apt.17734. Epub 2023 Oct 2. PMID 37786277
- [Derived] Harrison SA, Bashir M, Moussa SE, McCarty K, Pablo Frias J, Taub R, Alkhouri N. Effects of Resmetirom on Noninvasive Endpoints in a 36-Week Phase 2 Active Treatment Extension Study in Patients With NASH. Hepatol Commun. 2021 Jan 4;5(4):573-588. doi: 10.1002/hep4.1657. eCollection 2021 Apr. PMID 33860116